CLINICAL TRIAL: NCT02480374
Title: A Phase I Study of the Safety and Biological Activity of Intraperitoneal IMNN-001 (IL-12 Plasmid Formulated with PEG-PEI-Cholesterol Lipopolymer) Administered in Combination with Standard Neoadjuvant Chemotherapy in Patients Newly Diagnosed with Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Study of Safety & Biological Activity of IP IMNN-001 (also Known As GEN-1) with Neoadjuvant Chemo in Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-14-101
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: GEN-1; IMNN-001
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — GEN-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Carboplatin + Paclitaxel + IMNN-001
  Interventions: Biological: IMNN-001

INTERVENTIONS:
Biological: IMNN-001
  Other Names: GEN-1

SUMMARY:
This dose escalation study will determine a maximum tolerated dose and/or optimal biological dose of GEN-1 for carboplatin/paclitaxel combination in newly diagnosed ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma per pre-treatment biopsies by laparoscopy, or interventional radiology or CT guided core biopsy. Histologic documentation of the original primary tumor is required via the pathology report.
2. Patients with the following histologic epithelial cell types are eligible: High grade serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified (N.O.S.).
3. Patients must have adequate:

   i. Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl. This ANC cannot have been induced or supported by granulocyte colony stimulating factors. Platelets greater than or equal to 100,000/mcl.

   ii. Renal function: Creatinine ≤ 1.5 x institutional upper limit normal (ULN). iii. Hepatic function: Bilirubin ≤ 1.5 x ULN. SGOT (AST) and SGPT (ALT) ≤ 3.0 x ULN and alkaline phosphatase ≤ 2.5 x ULN.

   iv. Neurologic function: Neuropathy (sensory and motor) less than or equal to Grade 1.
4. Patients should be free of active infection requiring parenteral antibiotics or a serious uncontrolled medical illness or disorder within four weeks of study entry.
5. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to the first treatment. Continuation of hormone replacement therapy is permitted.
6. Patients must have a performance status score of 0, 1 or 2 by Eastern Cooperative Group (ECOG) criteria.
7. Patients of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of protocol therapy and be practicing an effective form of contraception. If applicable, patients must discontinue breastfeeding prior to study entry.
8. Patients must have satisfactory results for the baseline laboratory analyses and diagnostic procedures as specified in the protocol.
9. Patients must have signed an IRB-approved informed consent and authorization permitting release of personal health information.
10. Patients must be at least 18 years old.

Exclusion Criteria:

1. Patients who have received prior treatment with IMNN-001.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to GEN-1 or other agents used in this study.
3. Patients who have received oral or parenteral corticosteroids within 2 weeks of study entry or who have a clinical requirement for ongoing systemic immunosuppressive therapy not related to chemotherapy administration.
4. Patients receiving treatment for active autoimmune disease. "Active" refers to any condition currently requiring therapy. Examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.
5. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted in the protocol are excluded if there is any evidence of other malignancy being present within the last three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
6. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
7. Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
8. Patients with known active hepatitis.
9. Patients with concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy.
10. Patients of childbearing potential, not practicing adequate contraception, patients who are pregnant, or patients who are breastfeeding are not eligible for this trial.
11. Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
12. Patients with any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration including: abdominal surgery within 4 weeks of study entry (for reasons other than IP port placement), intestinal dysfunction, or suspected extensive adhesions from prior history or finding at laparoscopy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
DLT | 4 weeks
  Dose-limiting toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Premal Thaker, M.D., Study Chair — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of Alabama Birmingham Cancer Center, Birmingham, Alabama
  - Washington Univ. in St. Louis/Barnes Jewish Hospital, St Louis, Missouri
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yin X, Davi R, Lamont EB, Thaker PH, Bradley WH, Leath CA 3rd, Moore KM, Anwer K, Musso L, Borys N. Historic Clinical Trial External Control Arm Provides Actionable GEN-1 Efficacy Estimate Before a Randomized Trial. JCO Clin Cancer Inform. 2023 Jan;7:e2200103. doi: 10.1200/CCI.22.00103. PMID 36608308
- [Derived] Gonzalez-Junca A, Liu FD, Nagaraja AS, Mullenix A, Lee CT, Gordley RM, Frimannsson DO, Maller O, Garrison BS, Iyer D, Benabbas A, Truong TA, Quach A, Tian M, Martinez R, Savur R, Perry-McNamara A, Nguyen D, Almudhfar N, Blanco C, Huynh C, Nand A, Lay YE, Magal A, Mangalampalli S, Lee PJ, Lu TK, Lee G. SENTI-101, a Preparation of Mesenchymal Stromal Cells Engineered to Express IL12 and IL21, Induces Localized and Durable Antitumor Immunity in Preclinical Models of Peritoneal Solid Tumors. Mol Cancer Ther. 2021 Sep;20(9):1508-1520. doi: 10.1158/1535-7163.MCT-21-0030. Epub 2021 Jul 1. PMID 34210826